CLINICAL TRIAL: NCT02573636
Title: The Predictive Value of Coexisting TMPRSS2-ERG Gene Fusion and PTEN Deletion in Prostate Cancer Patients with Biochemical Failure Status Post Salvage or Radical Radiation Therapy
Status: Recruiting | Type: Observational
Sponsor: Sir Mortimer B. Davis - Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Dr. Tamim Niazi, Principal investigator, Sir Mortimer B. Davis - Jewish General Hospital
Other Study IDs: PCS VIII
Record Dates: First submitted 2015-10-05; First posted 2015-10-12 (Estimated); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Areas of prostate tumor will be identified by the pathologist of the study. This will then be excised from the paraffin block using a tissue microarray punch. Two punches will be acquired: one for RNA extraction and one for DNA extraction. RNA and DNA will be extracted using the RecoverAll Nucleic Acid Isolation Kit (Ambion). Standard protocol for the isolation of nucleic acids will be used differing only in the time of protease digestion such that RNA is isolated after a short incubation (30 minutes), while DNA is isolated after a longer incubation (overnight). DNA will be used to assess copy number variation at the PTEN locus (10q23) using quantitative PCR and appropriate Taqman chemistry.
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of the study is to evaluate the predictive value of TMPRSS2-ERG gene fusion and PTEN in patients with high risk prostate cancer treated with first line LHRH agonist after biochemical failure.

DETAILED DESCRIPTION:
The objective of the study is to evaluate the predictive value of TMPRSS2-ERG gene fusion and PTEN in patients with high risk prostate cancer treated with first line LHRH agonist after biochemical failure.

Patients in this study will be treated with standard hormonal treatment. Patients will remain on treatment regardless of rising PSA. PSA, other systemic therapy maybe added and the patients with oligometastasis could be treated with radiation therapy; this would be at the discretion of the treating oncologist.

The primary endpoint of this study is to determine the predictive value of TMPRSS2-ERG gene fusion and PTEN in hormonal refractory free survival and clinical progression rate in three years. The secondary endpoints are to evaluate the relation between Gleason score and TMPRSS2-ERG gene fusion and PTEN independently and together, the relation between T stage and TMPRSS2-ERG gene fusion and PTEN independently and together, and to determine the association of these markers with overall survival.

ELIGIBILITY:
Inclusion Criteria:

* T3a +
* PSA > 20
* Gleason 8 or higher
* Karnofsky performance status ≥ 70.
* Signed study-specific informed consent

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The original slides of 208 patients with informed consent will be reviewed. Patients with and without markers under the investigation will be accrued into this study. The investigators at the treating institutions will submit paraffin-embedded tissue blocks from the original pre-treatment diagnostic prostatic biopsy, which will be reviewed to confirm the Gleason score and to record other histopathologic features, such as the extent of tumor in the biopsies, the number of positive biopsies, and mitotic index.
Sampling Method: Non-Probability Sample
Enrollment: 208 (Estimated)
Dates: Start 2016-03 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Number of patients with biochemical failure showing coexistence of PTEN and TMPRSS2-ERG gene fusion. | recruitment over 4 years
  Biopsy samples of patients treated for high risk prostate cancer with radical radiation and hormonal therapy (LHRH) who have either clinical progression or 3-year hormonal refractory free survival will be tested to evaluate the predictive value of the coexistence of TMPRSS2-ERG gene fusion and the PTEN deletion. The results between the two groups will be compared to see if either DNA changes are an indicator of LHRH refractoriness

CONTACTS AND LOCATIONS:
Locations (9):
- Canada (9):
  - CIUSSS du Saguenay-Lac-St-Jean/CSSS de Chicoutimi, Chicoutimi, Quebec
  - CISSS de la Montérégie-Centre - Hôpital Charles-LeMoyne, Greenfield Park, Quebec
  - CISSS de Laval - Hôpital de la Cité-de-la-santé de Laval, Laval, Quebec
  - CIUSSS de l'Est-de-l'Île-de-Montréal - Hôpital Maisonneuve-Rosemont, Montreal, Quebec
  - Jewish General Hospital, McGill University, Montreal, Quebec
  - MUHC - Cedars Cancer Center, Montreal, Quebec
  - CHU - L'Hôtel-Dieu de Québec, Québec, Quebec
  - CIUSSS de l'Estrie - Hôpital Fleurimont, Sherbrooke, Quebec
  - CIUSSS de la Mauricie-et-du-centre-du Quebec - Centre hospitalier régional de Trois-Rivières, Trois-Rivières, Quebec

IPD SHARING:
Plan to Share IPD: No